CLINICAL TRIAL: NCT06784830
Title: Enhancing Nursing Interventions for Alzheimer's Patients During PET/CT Imaging: Effects on Image Quality and Patient Satisfaction
Brief Title: Nursing Interventions for Alzheimer's Patients During PET/CT Imaging
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sichuan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Hao Wang, Associate senior physician, Sichuan Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SichuanPPH-HL
Record Dates: First submitted 2025-01-09; First posted 2025-01-20 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-01

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Refinement of specialized nursing intervention (Experimental): This specialized nursing emphasizes individualized care plans customized to each patient's unique condition, targeting improvements in both the treatment experience and overall results.
  Interventions: Other: Effects on Image Quality and Patient Satisfaction; Other: Anxiety degree of patients after nursing
- Routine nursing intervention (No Intervention): The nurse gave pre-examination education to the control group. All the subjects rested in the waiting room and waited for examination. During the examination, the examination was completed according to the general nursing measures corresponding to different tracers.

INTERVENTIONS:
Other: Effects on Image Quality and Patient Satisfaction — Effect of nursing intervention on image quality and patient satisfaction during PET/CT imaging in Alzheimer's patients
  Arms: Refinement of specialized nursing intervention
Other: Anxiety degree of patients after nursing — Self Rating Anxiety will be used Scale (SAS) to assess the degree of anxiety after care
  Arms: Refinement of specialized nursing intervention

SUMMARY:
The impact of nursing Interventions during PET/CT imaging in Alzheimer's patients on image quality and patient satisfaction will be assessed in 200 patients.

DETAILED DESCRIPTION:
This study will analyze clinical data from 200 Alzheimer's disease (AD) patients who underwent PET imaging and were admitted to Sichuan Provincial People's Hospital over a period of six months. The control group will receive routine nursing intervention, while the observation group will receive a refined specialized nursing intervention. We will meticulously compare various performance aspects in both groups to assess the impact of refined specialized nursing intervention on patients' image quality and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Meet the criteria for diagnosing dementia as described in the fourth edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV-R), Use the diagnostic criteria for AD from the National Institute of Neurology, Speech and Communication Disorders and Stroke - Alzheimer's Disease and Related Disorders (NINCDS-ADRDA) or the National Institute on Aging and Alzheimer's Disease Association (NIA-AA).

Exclusion Criteria:

* Patients with a history of stroke and focal neurological signs, and imaging findings consistent with small cerebral vascular disease (Fazekas score ≥2);
* The presence of other neurological disorders that can cause brain dysfunction (e.g., depression, brain tumors, Parkinson's disease, metabolic encephalopathy, encephalitis, multiple sclerosis, epilepsy, brain trauma, Normal facial pressure hydrocephalus);
* The presence of other systemic diseases that can cause cognitive impairment (such as liver insufficiency, renal insufficiency, thyroid dysfunction, severe anemia, folic acid or vitamin B12 deficiency, syphilis, HIV infection, alcohol and drug abuse, etc.);
* There is mental and neurological retardation.
* There are other diseases that are known to cause cognitive impairment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-06-15 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-02-20 (Estimated)

PRIMARY OUTCOMES:
Comparison of refined nursing and routine nursing intervention in Alzheimer's Patients during PET/CT Imaging | through study completion, an average of 6 months
  The control group received routine care. The nurse gave pre-examination education to the control group, and all the subjects rested in the waiting room and waited for examination. During the examination, the examination was completed according to the general nursing measures corresponding to different tracers, and the examination was completed by leaving the examination room after the end. The patients in the observation group were educated before examination and received refined nursing measures on the basis of routine nursing.

CONTACTS AND LOCATIONS:
Overall Officials: Hao Wang, Doctor, Study Director — Sichuan Provincial People's Hospital
Locations (1):
- Departments of Nuclear Medicine, Sichuan Provincial People's Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No